CLINICAL TRIAL: NCT03793790
Title: Learning Mechanisms in Nocebo Hyperalgesia: the Role of Conditioning and Extinction Processes
Brief Title: The Role of Learning in Nocebo Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Universiteit Leiden (Other)
Responsible Party: Principal Investigator, AWMEvers, Prof. Dr., Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CEP18-0816/318
Record Dates: First submitted 2018-12-29; First posted 2019-01-04 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Nocebo Effects; Hyperalgesia; Chronic Pain; Pain Syndrome
Keywords: Nocebo; Pain; Conditioning; Counterconditioning; Partial reinforcement; Learning
MeSH Terms: conditions — Hyperalgesia; Chronic Pain; Somatoform Disorders; Pain | interventions — Extinction, Biological

STUDY DESIGN:
Intervention Model Description: This study employs a 2-by-2 design (i.e.,2 conditioning induction groups and 2 attenuation groups), with an additional control group (i.e., sham conditioning). Participants are thus allocated in 1 out of 5 groups.
Who Masked: Participant, Investigator
Masking Description: A double-blind randomization list (stratified for gender) was created by an independent statistician. Complete blinding of the researchers during the experiment is not possible due to the nature of conditioning paradigms. However, in this study blinding is optimized: the researchers are informed of the (conditioning) group to which participants are allocated after their final inclusion to the study, and after all questionnaires and pain calibration procedures have been completed on the testing day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Conditioning nocebo effects on pain with a partial reinforcement schedule (induction) and counterconditioning of the previously induced nocebo effect (attenuation).
  Interventions: Behavioral: Conditioning with partial reinforcement; Behavioral: Counterconditioning
- Group 2 (Experimental): Conditioning nocebo effects on pain with a partial reinforcement schedule (induction) and extinction of the previously induced nocebo effect (attenuation).
  Interventions: Behavioral: Conditioning with partial reinforcement; Behavioral: Extinction
- Group 3 (Experimental): Conditioning nocebo effects on pain with a continuous reinforcement schedule (induction) and counterconditioning of the previously induced nocebo effect (attenuation).
  Interventions: Behavioral: Conditioning with continuous reinforcement; Behavioral: Counterconditioning
- Group 4 (Experimental): Conditioning nocebo effects on pain with a continuous reinforcement schedule (induction) and extinction of the previously induced nocebo effect (attenuation).
  Interventions: Behavioral: Conditioning with continuous reinforcement; Behavioral: Extinction
- Group 5 (Sham Comparator): Sham conditioning of nocebo effects on pain (induction) and extinction (attenuation).
  Interventions: Behavioral: Sham Conditioning

INTERVENTIONS:
Behavioral: Conditioning with partial reinforcement — Conditioning with partial reinforcement (PRF) provides an uncertain pairing of unconditioned high pain stimuli and conditioned stimuli (i.e., on-screen messages signaling the activation of a mock medical device). During PRF only 70 percent of unconditioned stimuli are paired to conditioned stimuli. Pain of only moderate intensity is used for control stimuli that are paired to the deactivation of the mock device and are also used in the 30 percent of unreinforced trials.
  Arms: Group 1; Group 2
Behavioral: Conditioning with continuous reinforcement — During conditioning with continuous reinforcement (CRF) unconditioned high pain stimuli are paired to conditioned stimuli (i.e., on-screen messages signaling the activation of a mock medical device) in 100 percent of conditioning trials. Pain of only moderate intensity is used for control stimuli that are paired to the deactivation of the mock device.
  Arms: Group 3; Group 4
Behavioral: Counterconditioning — During counterconditioning, the previously conditioned nocebo effects on pain are attenuated by pairing the same conditioned stimuli (i.e., on-screen messages signaling the activation of a mock medical device) to thermal pain stimuli of low intensity.
  Arms: Group 1; Group 3
Behavioral: Extinction — During extinction, the previously conditioned nocebo effects on pain are attenuated by pairing the same conditioned stimuli (i.e., on-screen messages signaling the activation of a mock medical device) only to control stimuli of moderate intensity (previously paired to the deactivation of the mock device).
  Arms: Group 2; Group 4
Behavioral: Sham Conditioning — In the sham group, participants receive different instructions (namely, that the activation of the device is not expected to affect their pain sensitivity). Additionally, during sham conditioning unconditioned stimuli are not consistently paired to conditioned stimuli, thereby preventing the formation of an association between high pain stimuli and the activation of the mock medical device. In the attenuation phase participants undergo an extinction procedure.
  Arms: Group 5

SUMMARY:
Nocebo effects are adverse effects induced by patients' expectations. Nocebo effects on pain may underlie several clinical conditions, such as chronic pain. These effects can be learned via classical conditioning mechanisms. In the lab, nocebo effects are commonly studied via conditioning with continuous reinforcement (CRF) during which 100 percent of unconditioned pain stimuli are paired to conditioned stimuli (i.e., the activation of a mock medical device). Partial reinforcement (PRF) provides a more uncertain pairing during conditioning, where less than 100 percent of unconditioned pain stimuli are paired to conditioned stimuli. This method provides a potentially more clinically relevant learning platform to study how nocebo effects on pain are induced. In this study, the efficacy of conditioning with PRF, CRF, and sham-conditioning in inducing nocebo effects on pain will be compared. Furthermore, a counterconditioning method will be compared to an extinction method for the attenuation of nocebo effects on pain. Given the relevance of nocebo effects for patients, it is important to ascertain effective & clinically relevant methods to understand how nocebo effects may be formed and attenuated. This study is conducted by Leiden University.

DETAILED DESCRIPTION:
Main planned analyses:

Primary Outcome; Comparing the effectivity of conditioning with PRF, conditioning with CRF, and sham conditioning, in inducing nocebo effects on pain:

The magnitude of the induced nocebo effect during the first evocation phase (dependent variable), will be compared between induction groups (independent variable). The pain ratings for the first control trial will be measured against the pain ratings for the first reinforced trial, yielding the magnitude of the nocebo effect. A 3x2 mixed model Analysis of Variance (ANOVA) will be used, treating group as the between-subjects factor with three levels (PRF, CRF, sham) and magnitude of the nocebo effect on pain as a within-subjects measure with two levels (first control and first reinforced trial). Planned contrasts will be conducted.

Secondary Outcome; Comparing the effectivity of counterconditioning and extinction in attenuating nocebo effects on pain:

The nocebo effect still present in the second evocation phase (dependent variable) will be compared between attenuation groups (independent variable). This effect will be measured as the change in pain ratings reported in the first reinforced trial of the first evocation phase (after induction) and pain ratings reported in the first reinforced trial of the second evocation phase (after attenuation). This effect will be further analysed by measuring any change in pain reports for the control trials (second dependent variable) in the same way. The effect of induction group will also be further explored. A 2x2 mixed model ANOVA will be conducted, with attenuation group as the between-subjects factor (counterconditioning and extinction) and the degree to which the nocebo effect has been attenuated as the within-subjects measure with two levels (first and second evocation phase for the first reinforced trials). Further secondary analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 35 years
* Good understanding of the Dutch language

Exclusion Criteria:

* Severe or chronic physical morbidity (e.g., heart and lung diseases, diabetes)
* Psychiatric disorders (DSM diagnosis; e.g., depression, autism)
* Chronic pain complaints (≥ 6 months) at present or in the past
* Current pain
* Current use of analgesic medication
* Pregnancy
* After inclusion, participants who do not reach a sensation of high pain with the highest temperature administered or participants who appear unable to distinguish between moderate and high pain stimuli will also be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants whose gender identity, gender expression, and lived gender is male, will be included as male. Participants whose gender identity, gender expression, and lived gender is female, will be included as female.
Enrollment: 140 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Magnitude of nocebo effects on pain (rated on a 0-10 numeric rating scale) after PRF, CRF, or sham conditioning. | Testing day 1, in the 1st evocation phase
  This will be calculated in the first evocation phase, by analysing the pain ratings for the first reinforced trial against the pain ratings for the first control trial.

SECONDARY OUTCOMES:
Magnitude of nocebo effects on pain (rated on a 0-10 numeric rating scale) still present after counterconditioning or extinction. | Testing day 1, in the 2nd evocation phase
  This will be calculated by analysing the pain ratings for the first reinforced trial in the second evocation phase against the pain ratings for the first reinforced trial in the first evocation phase.

OTHER OUTCOMES:
Possible resistance to extinction of induced nocebo effects on pain (rated on a 0-10 numeric rating scale) after PRF as compared to after CRF. | Testing day 1, in the attenuation phase and the 2nd evocation phase
  Exploring whether participants in the PRF group will exhibit higher resistance to extinction during attenuation, as compared to participants in the CRF group. This will be assessed by analyzing the time-course of extinction of the previously induced nocebo effects on pain (rated on a 0-10 numeric rating scale) during the attenuation phase and the 2nd evocation phase

CONTACTS AND LOCATIONS:
Overall Officials: Andrea WM Evers, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data are collected pseudonymised thus no personal data are stored or shared. Consent forms are the only sources containing personal data and will not be shared, but are monitored by the department's Data Monitor.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available immediately after publication of the study and will be retained for 15 years.
Access Criteria: Data can be shared with scientists in relevant fields for the purpose of future studies such as replication or meta-analysis (or with designated persons for monitoring purposes).